CLINICAL TRIAL: NCT02265354
Title: Developing Smokers for Smoker (S4S): A Collective Intelligence Tailoring System
Acronym: S4S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Massachusetts, Amherst (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rajani Sadasivam, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H00002005; K07CA172677 (NIH)
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Tobacco Smoking
Keywords: Tobacco Smoking Cessation; Computer tailored health communication; messaging; collective intelligence; recommender systems; machine learning
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collective-Intelligence computer tailored health communication (Experimental): Smokers will have access to all Decide2quit.org website functions and will receive 4 tailored emails per week based on a collective intelligence recommender systems algorithm for up to 6 months
  Interventions: Behavioral: Collective-Intelligence computer tailored health communication
- Rule-based computer tailored health communication (Active Comparator): Smokers will have access to all Decide2quit.org website functions and will receive 4 tailored emails per week based on a rule-based algorithm for up to 6 months
  Interventions: Behavioral: Rule-based computer tailored health communication

INTERVENTIONS:
Behavioral: Collective-Intelligence computer tailored health communication
  Arms: Collective-Intelligence computer tailored health communication
Behavioral: Rule-based computer tailored health communication
  Arms: Rule-based computer tailored health communication

SUMMARY:
This study will advance computer tailoring by adapting machine learning collective intelligence algorithms that have been used outside healthcare by companies like Amazon and Google to enhance the personal relevance of the health communication.

DETAILED DESCRIPTION:
Smoking is still the number one preventable cause of cancer death. New approaches are needed to engage smokers in the 21st century in smoking cessation. I propose to develop S4S (Smokers for Smoker), a next-generation patient-centered computer tailored health communication (CTHC) system. Unlike current rule-based CTHCs, S4S will replace rules with complex machine learning algorithms, and use the collective experiences of thousands of smokers engaged in a web-assisted tobacco intervention to enhance personally-relevant tailoring for new smokers entering the system. The investigators will adapt collective intelligence algorithms that have been used outside healthcare by companies like Amazon and Google to enhance CTHC. Using knowledge from scientific experts, current CTHC collect baseline patient "profiles" and then use expert-written, rule-based systems to tailor messages to patient subsets. Such theory-based "market segmentation has been effective in helping patients reach lifestyle goals. However, there is a natural limit in the ability of a rule-based system to truly personalize content, and adapt personalization over time. Current CTHC have reached this limit, and the investigators propose to go beyond. The investigators first aim is to develop the Web 2.0 "S4S" recommender system. The investigators second aim is to evaluate S4S within the context of a NCI funded web-assisted tobacco intervention (Decide2Quit.org).

ELIGIBILITY:
Inclusion Criteria:

* Current Smokers

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Repeated Use of website measure | Every Login for 6 months
  This measure is an ordinal scale of the number of functions used after the first visit to the Decide2Quit.org website (0: use of no functions, 1: use of 1-2 functions, 2: use of 2-4 functions, see Table 9 list of functions). We will use scripts on the website to assess this information

SECONDARY OUTCOMES:
30-day point prevalent smoking cessation at six months | At 6 months
  Did you smoke any cigarettes during the past 30 days? This will be assessed using a follow-up Telephone or Internet survey

CONTACTS AND LOCATIONS:
Overall Officials: Rajani S Sadasivam, PhD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States